CLINICAL TRIAL: NCT03185325
Title: Micro Ribosomal Nucleic Acid 155 in Non Hodgkin Lymphoma
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Merna Narouz, principal investigator, Assiut University
Other Study IDs: AssiutUniversity
Record Dates: First submitted 2017-06-10; First posted 2017-06-14 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-01

CONDITIONS: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood and bone marrow samples for micro ribonucleic acid 155 extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non hodgkin lymphoma patients: bone marrow puncture and venous blood samples
  Interventions: Other: bone marrow puncture and venous blood samples
- healthy voulnteers: venous blood samples
  Interventions: Other: venous blood samples

INTERVENTIONS:
Other: bone marrow puncture and venous blood samples — bone marrow and peripheral blood samples are collected in non hodgkin lymphoma patients
  Groups: Non hodgkin lymphoma patients
Other: venous blood samples — venous blood samples are collected in healthy voulnteers
  Groups: healthy voulnteers

SUMMARY:
Lymphomas are hematological malignancies, which are divided into non-Hodgkin lymphoma and Hodgkin lymphoma. Non hodgkin lymphoma is a lymphoma-derived malignancy that makes up about 90% of all malignant lymphoma. According to its origin, non hodgkin lymphoma is classified into B-cell non hodgkin lymphoma and T-cell non hodgkin lymphoma. The most common types are follicular lymphoma, and diffuse large B-cell lymphoma. Lymphomas are types of cancer that develops from lymphocytes, a type of white blood cell. Diagnosis is by examination of a bone marrow or lymph node biopsy. Non hodgkin lymphoma mortality has increased in recent years and has become the seventh most frequently occurring cancer.

DETAILED DESCRIPTION:
Biomarkers are defined as objective indicators of biological processes, pathogenic processes, or pharmacological response to a therapeutic intervention. Diagnostic biomarkers which are type of biomarkers, identify the presence of disease, differentiate normal from malignant, distinguish different diagnoses or progression stages.

Micro ribosomal nucleic acids have been demonstrated to possess biomarker potentiality in multiple diseases, both individually and when combined in signature profiles. Micro ribosomal nucleic acids are short single-stranded noncoding ribosomal nucleic acids of 20-22 nucleotides that function to regulate gene expression at the posttranscriptional level. They play fundamental roles in the regulation of cellular proliferation, differentiation, and apoptosis. Dysregulation of micro ribosomal nucleic acid is a unique feature of cancers including lymphomas . Information about the functional role of micro ribosomal nucleic acid dysregulation in lymphomas is increasing day by day.

The present study focuses on the micro ribosomal nucleic acid 155 since this molecule represents a typical multifunctional micro ribosomal nucleic acid. To date, increased evidence points out that micro ribosomal nucleic acid 155 is involved in numerous biological processes including haematopoiesis, inflammation and immunity. Deregulation of micro ribosomal nucleic acid 155 has been found to be associated with different kinds of cancer, cardiovascular diseases and viral infections. Since investigation on the functional activity of micro ribosomal nucleic acid 155 started a few years ago, it is reasonable to predict that many other functions will be uncovered in the near future.

Micro ribosomal nucleic acid 155 maps within and is processed from an exon of a noncoding ribosomal nucleic acid transcribed from the B-cell Integration Cluster located on chromosome 21.

Micro ribosomal nucleic acid 155 is an oncological micro ribosomal nucleic acid with a crucial role in tumor initiation and development of several B-cell malignancies. Micro ribosomal nucleic acid 155 was upregulated in several malignancies compared to nonmalignant controls and overexpression of micro ribosomal nucleic acid 155 was further associated with poor prognosis. Elevated expression of micro ribosomal nucleic acid 155 shows potentiality as a diagnostic and prognostic biomarker in diffuse large B-cell lymphoma and chronic lymphocytic leukemia. Additionally, in vitro and in vivo studies suggest micro ribosomal nucleic acid 155 as an efficient therapeutic target, supporting its oncogenic function. The use of inhibiting anti-micro ribosomal nucleic acid structures indicates promising potential as novel anticancer therapeutics.

The search for non-invasive tools for the diagnosis and management of cancer has long been a goal of cancer research that has led to great interest in the field of circulating nucleic acids in plasma and serum.

ELIGIBILITY:
Inclusion Criteria:

* Non hodgkin lymphoma patients of any age or sex.
* healthy volunteers within the same range of age.

Exclusion Criteria:

* patients with any other haematological malignancy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Non hodgkin lymphoma patients who are newly diagnosed or relapsed cases and healthy controls who have no other heamatological malignancies
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
mean difference of micro ribosomal nucleic acid 155 expression levels between samples of both non hodgkin lymphoma patients and healthy controls | 6 months
  measuring levels of micro ribosomal nucleic acid 155 in peripheral blood and bone marrow samples of non hodgkin lymphoma patients and in peripheral blood samples of healthy controls

SECONDARY OUTCOMES:
Mean difference of levels of expression of micro ribosomal nucleic acid 155 between peripheral blood and bone marrow samples of non hodgkin lymphoma patients | 6 months
  measuring levels of expression of micro ribosomal nucleic acid 155 in peripheral blood and bone marrow samples in non hodgkin lymphoma patients

CONTACTS AND LOCATIONS:
Overall Officials: Merna W Narouz, Principal Investigator — Assiut University
Locations (1):
- AssiutU, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ekstrom-Smedby K. Epidemiology and etiology of non-Hodgkin lymphoma--a review. Acta Oncol. 2006;45(3):258-71. doi: 10.1080/02841860500531682. PMID 16644568
- [Background] Nogai H, Dorken B, Lenz G. Pathogenesis of non-Hodgkin's lymphoma. J Clin Oncol. 2011 May 10;29(14):1803-11. doi: 10.1200/JCO.2010.33.3252. Epub 2011 Apr 11. PMID 21483013
- [Background] Willis TG, Dyer MJ. The role of immunoglobulin translocations in the pathogenesis of B-cell malignancies. Blood. 2000 Aug 1;96(3):808-22. No abstract available. PMID 10910891
- [Background] Jansson MD, Lund AH. MicroRNA and cancer. Mol Oncol. 2012 Dec;6(6):590-610. doi: 10.1016/j.molonc.2012.09.006. Epub 2012 Oct 9. PMID 23102669